CLINICAL TRIAL: NCT02607592
Title: Nedaplatin or Cisplatin Combined With Pemetrexed in the First Line Treatment of Advanced Adenocarcinoma：A Prospective Multi-center Phase III Randomized Controlled Trial
Brief Title: A Prospective Multi-center Phase III Randomized Controlled Trial
Acronym: NACA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, associate professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201507003
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma，Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung cancer; overall toxicity value
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nedaplatin and Pemetrexed (Experimental): nedaplatin 90mg/m2 d1+pemetrexed 500mg/m2 d1 （Every three weeks for a treatment cycle）
  Interventions: Drug: nedaplatin+pemetrexed
- Cisplatin and Pemetrexed (Active Comparator): cisplatin 25mg/m2 d1-3+pemetrexed 500mg/m2 d1 （Every three weeks for a treatment cycle）
  Interventions: Drug: cisplatin and pemetrexed

INTERVENTIONS:
Drug: cisplatin and pemetrexed — cisplatin 25mg/m2 d1-3+pemetrexed 500mg/m2 d1 （Every three weeks for a treatment cycle）
  Arms: Cisplatin and Pemetrexed
Drug: nedaplatin+pemetrexed — nedaplatin 90mg/m2 d1+pemetrexed 500mg/m2 d1 （Every three weeks for a treatment cycle）
  Arms: Nedaplatin and Pemetrexed

SUMMARY:
The purpose of this study is to investigate the PFS, ORR, OS and overall toxicity value（OTV）on advanced adenocarcinoma treated with nedaplatin or cisplatin combined with pemetrexed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who was confirmed primary adenocarcinoma by pathologic histology or cytology
2. The TNM staging system according to IASLC2009 was stageIV or those stageIIIB who were not fit for operation or radiotherapy
3. Including one available evaluation lesion at least according to RECIST criteria
4. Adult patients (≥18 years and ≤75 years). ECOG Performance Status 0 or 1 .Life expectancy of at least 12 weeks.Haemoglobin ≥90g/dl, Absolute neutrophil count (ANC)≥ 2x 109/L, platelets ≥100 x 109/L. Total bilirubin ≤upper limit of normal (ULN). ALT and AST ≤ 2.5 x ULN. Creatinine clearance ≥60ml/min (calculated according to Cockcroft-gault formula).
5. Patients who had never received any antineoplastic therapy

Exclusion Criteria:

1. Patient who has another cancer in recent 5 years,not including basal cell carcinoma or cervical carcinoma in situ
2. Patient with brain metastases whose intracranial pressure symptoms can not control by using glucocorticoid or mannitol
3. Previous radiotherapy（Palliative radiotherapy in order to pain management can be excluded）
4. Patient who has used chemotherapy before(bisphosphonate can be excluded )
5. Serious uncontrolled systemic disease including active infection,uncontrolled hypertension,diabetes,unstable angina,congestive heart failure,myocardial infarction,severe arrhythmia which needs drugs,hepatic、renal and metabolic disease
6. Patient who is allergic to drugs we need to use
7. Patients who are in pregnancy or lactation
8. AST or ALT 》2.5 * upper limit of normal (ULN)，and ALP》5*ULN

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Estimated)
Dates: Start 2015-08; Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
progression free-survival（PFS） | 12months
  Progression-free survival is defined as the time from the starting date of study drug to the date of first documentation of disease progression or death, whichever occurs first

SECONDARY OUTCOMES:
objective response rate （ORR） | 12months
  ORR is defined as the proportion (%) of patients with at least one visit response of complete response (CR) or partial response (PR).
overall survival（OS） | 24 months
  OS is defined as the time from the starting date of study drug to the date of death due to any cause
overall toxicity value | 12 months
  toxicity graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0
Progression-Free Survival (PFS) rate at 18 weeks | 20 weeks
  the proportion (%) of patients without disease progression at 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: li-kun Chen, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University of cancer center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Pfister DG, Johnson DH, Azzoli CG, Sause W, Smith TJ, Baker S Jr, Olak J, Stover D, Strawn JR, Turrisi AT, Somerfield MR; American Society of Clinical Oncology. American Society of Clinical Oncology treatment of unresectable non-small-cell lung cancer guideline: update 2003. J Clin Oncol. 2004 Jan 15;22(2):330-53. doi: 10.1200/JCO.2004.09.053. Epub 2003 Dec 22. No abstract available. PMID 14691125